CLINICAL TRIAL: NCT02928744
Title: Evaluation of the Reversibility of the Bronchial Obstruction by Impulse Oscillometry Technique in Chronic Obstructive Pulmonary Disease (COPD): Correlation With Functional Features Measured by Plethysmography and Dyspnoea
Acronym: OSCILLOREVERS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/43; 2011-A00964-37 (Other: AFSSAPS)
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: COPD
Keywords: Resistance; Forced oscillations; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD (Experimental)
  Interventions: Other: COPD

INTERVENTIONS:
Other: COPD — Plethysmography
Other: COPD — Forced oscillations

SUMMARY:
Limitation of expiratory flows is considered as the main determiner of dynamic distension and dyspnoea in chronic obstructive pulmonary disease (COPD). The analysis of proximal and distal resistances should allow to better appreciate the functional impact.

This study should also allow to specify the best parameters in respiratory functional explorations useful for the follow-up in COPD and to specify the relevance of functional indications other than the forced expiration volume at 1 second (FEV1) or the functional residual capacity (FRC) to estimate in a more relevant way the clinical improve with the increase of the therapeutic load (increase of posology, association of two bronchodilatators, addition of an anti-inflammatory drug, thus etc…) at already handled patients suffering from a persistent dyspnoea insufficiently relieved.

ELIGIBILITY:
Inclusion Criteria:

* COPD with dyspnoea with Medical Research Council scale (MRC) >1,
* No exacerbation for 6 weeks
* No bronchodilatator short action(share) (ß 2 agonist or ipratropium) within 6 hours before the respiratory evaluation and the test of reversibility.
* Patient under current treatment (ß2 long-acting agonist (LABA) or anticholinergic long-acting (LLAMA(LAMA)) or LABA-corticoid association inhaled (CSI), or triples LABA-CSI-LAMA association) stable for at least 4 weeks, and taken for at least the 1 hour the day of the visit
* Having given a written consent

Exclusion Criteria:

* Patient Under 18
* Other respiratory illness
* Clinically significant left cardiac failure
* Obesity with BMI > 35 kg / m2)
* Unable to perform respiratory evaluations
* Contraindication to the salbutamol or to the ipratropium bromide or to one of its components
* Pregnant or breast-feeding woman
* Unable to agree
* No social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentage of obstruction reversibility | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Neveu, Principal Investigator — Hôpital Foch
Locations (2):
- France (2):
  - CHRU, Lille
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Rouzic O, Picaud M, Salvator H, Bautin N, Devillier P, Perez T. Residual reversibility in COPD patients already on long-acting bronchodilator: The OscilloRevers Study. Respir Med Res. 2024 Jun;85:101082. doi: 10.1016/j.resmer.2023.101082. Epub 2024 Jan 26. PMID 38280281